CLINICAL TRIAL: NCT01335490
Title: Intervening to Improve Birth Weight and Infant Respiratory Health in Rural Ghana
Brief Title: Intervening to Improve Infant Health in Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Global Alliance for Clean Cookstoves (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAF3520; 1R01ES019547-01A1 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Very Low Birth Weight Baby; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Biolite Cook Stove (Experimental): Provision of two cook stoves to each subject. Each stove burns wood fuel, but more efficiently than a traditional three stone fire.
  Interventions: Other: Cook stoves, either Biolite wood stove, or liquified petroleum gas stove plus fuel
- LPG Cook Stove (Experimental): Provision of a two-burner liquified petroleum gas stove to each subject, along with fuel needed for the family during the follow up period.
  Interventions: Other: Cook stoves, either Biolite wood stove, or liquified petroleum gas stove plus fuel
- Control (No Intervention)

INTERVENTIONS:
Other: Cook stoves, either Biolite wood stove, or liquified petroleum gas stove plus fuel — The cooking stoves will reduce air emissions significantly in the home, resulting in improved infant health. It will be given to the mother in the second or third trimester.
  Arms: Biolite Cook Stove; LPG Cook Stove

SUMMARY:
The purpose of the study is to understand how cooking might affect the health of pregnant women and their babies.

The goal of the research is to determine whether, interventions in decreasing exposure to smoke from cook stoves can bring about a significant change in the indoor air pollution levels and health of communities in Ghana.

Hypothesis 1. Use of improved cook stoves starting by the third trimester pregnancy will lead to a significant increase in average birth weight in newborns.

Hypothesis 2. Use of improved cook stoves will lead to a significant reduction in the rate of severe acute lower respiratory disease during the first 12 months of life.

DETAILED DESCRIPTION:
2. Overview of design and analysis [per CONSORT 2010] 2.1 Trial design [CONSORT 3a] The study is a three-arm cluster randomized trial, with two intervention arms and a control arm. The primary justification for intervening at the village level is that an individual level randomization, which would entail treatments and controls living side-by-side in a village, could lead to conflict within villages.

2.2 Study Participants [CONSORT 4a, 4b] The study will take place in the catchment area of Kintampo Health Research Centre. This comprises a population of 146,000. The study population is primarily rural and agricultural, and cooks primarily with biomass fuels. The study area is well described in Owusu-Agyei et al. 2012 (38).

A cluster was eligible to participate if it:

* Is located in Kintampo North or South Districts (this is the core study area for KHRC)
* Is primarily rural (in practice, this excludes Kintampo, which is a small city of approximately 40,000 people);
* Is operationally feasible (in practice, this excluded a handful very small, isolated clusters that would have presented extraordinary logistical challenges);
* Is home to women who primarily deliver at one of our four staffed birth facilities (in practice this excluded one village on the edge of the study area, in which women travel to another district for deliveries).

A woman will be eligible to participate in the study if she:

* Is in the first or second trimester of pregnancy (gestational age ≤ 24 weeks gestation; this is to ensure that the intervention is actually delivered prior to 27 weeks)
* Is carrying a live singleton fetus (twins will be excluded)
* Is the primary cook in her household or compound; and
* Is a non-smoker. 2.3 Interventions [CONSORT 5]

The study has three arms:

1. LPG intervention arm, in which households receive a two burner LPG cookstove and monthly gas deliveries;
2. An efficient biomass arm, in which households receive two BioLite cookstoves; and
3. A control arm 2.4 Outcomes [CONSORT 6a]

The primary health outcome measures for the study are:

1. Infant weight at birth, and
2. Physician assessed pneumonia. Baseline assessments of outcomes No baseline data for ALRI prevalence from Ghana is available. Our study will thus provide very valuable baseline data regarding this important disease.

KHRC has, in the course of conducting other research projects, captured some information regarding birth weight; statistics calculated from these data were used as inputs into power calculations. These data are described in (39).

2.5 Sample size [CONSORT 7a, 7b] For the three-arm design, we calculate that we need to enroll households to achieve our target of 1225 births (assuming that 85% of the pregnancies will result in a recorded birth after, accounting for move out, drop out, and still birth rates). These will be spread across 35 or more clusters, as outlined in the following table.

Clusters Births Enrollment BioLite 13 455 525 Control 13 455 525 LPG 9 315 365 total 35 1225 1415

ELIGIBILITY:
A cluster was eligible to participate if it:

* Is located in Kintampo North or South Districts (this is the core study area for KHRC)
* Is primarily rural (in practice, this excludes Kintampo, which is a small city of approximately 40,000 people);
* Is operationally feasible (in practice, this excluded a handful very small, isolated clusters that would have presented extraordinary logistical challenges);
* Is home to women who primarily deliver at one of our four staffed birth facilities (in practice this excluded one village on the edge of the study area, in which women travel to another district for deliveries).

A woman will be eligible to participate in the study if she:

* Is in the first or second trimester of pregnancy (gestational age ≤ 24 weeks gestation; this is to ensure that the intervention is actually delivered prior to 27 weeks)
* Is carrying a live singleton fetus (twins will be excluded)
* Is the primary cook in her household or compound; and
* Is a non-smoker.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1414 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Low birth weight | Birth

SECONDARY OUTCOMES:
Acute lower respiratory disease | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kinney, ScD, Principal Investigator — Columbia University
Locations (2):
- Columbia University Medical Center, New York, New York, United States
- Kintampo Medical Research Center, Kintampo, Ghana

REFERENCES:
- [Derived] Agyapong PD, Jack D, Kaali S, Colicino E, Mujtaba MN, Chillrud SN, Osei M, Gennings C, Agyei O, Kinney PL, Kwarteng A, Perzanowski M, Dwommoh Prah RK, Tawiah T, Asante KP, Lee AG. Household Air Pollution and Child Lung Function: The Ghana Randomized Air Pollution and Health Study. Am J Respir Crit Care Med. 2024 Mar 15;209(6):716-726. doi: 10.1164/rccm.202303-0623OC. PMID 38016085
- [Derived] Boamah-Kaali E, Jack DW, Ae-Ngibise KA, Quinn A, Kaali S, Dubowski K, Oppong FB, Wylie BJ, Mujtaba MN, Gould CF, Gyaase S, Chillrud S, Owusu-Agyei S, Kinney PL, Asante KP, Lee AG. Prenatal and Postnatal Household Air Pollution Exposure and Infant Growth Trajectories: Evidence from a Rural Ghanaian Pregnancy Cohort. Environ Health Perspect. 2021 Nov;129(11):117009. doi: 10.1289/EHP8109. Epub 2021 Nov 29. PMID 34842444
- [Derived] Jack DW, Ae-Ngibise KA, Gould CF, Boamah-Kaali E, Lee AG, Mujtaba MN, Chillrud S, Kaali S, Quinn AK, Gyaase S, Oppong FB, Carrion D, Agyei O, Burkhart K, Ana-Aro JA, Liu X, Berko YA, Wylie BJ, Etego SA, Whyatt R, Owusu-Agyei S, Kinney P, Asante KP. A cluster randomised trial of cookstove interventions to improve infant health in Ghana. BMJ Glob Health. 2021 Aug;6(8):e005599. doi: 10.1136/bmjgh-2021-005599. PMID 34452940
- [Derived] Kinney PL, Asante KP, Lee AG, Ae-Ngibise KA, Burkart K, Boamah-Kaali E, Twumasi M, Gyaase S, Quinn A, Oppong FB, Wylie BJ, Kaali S, Chillrud S, Yawson A, Jack DW, Owusu-Agyei S. Prenatal and Postnatal Household Air Pollution Exposures and Pneumonia Risk: Evidence From the Ghana Randomized Air Pollution and Health Study. Chest. 2021 Nov;160(5):1634-1644. doi: 10.1016/j.chest.2021.06.080. Epub 2021 Jul 21. PMID 34298005
- [Derived] Ae-Ngibise KA, Wylie BJ, Boamah-Kaali E, Jack DW, Oppong FB, Chillrud SN, Gyaase S, Kaali S, Agyei O, Kinney PL, Mujtaba M, Wright RJ, Asante KP, Lee AG. Prenatal maternal stress and birth outcomes in rural Ghana: sex-specific associations. BMC Pregnancy Childbirth. 2019 Oct 29;19(1):391. doi: 10.1186/s12884-019-2535-9. PMID 31664941
- [Derived] Lee AG, Kaali S, Quinn A, Delimini R, Burkart K, Opoku-Mensah J, Wylie BJ, Yawson AK, Kinney PL, Ae-Ngibise KA, Chillrud S, Jack D, Asante KP. Prenatal Household Air Pollution Is Associated with Impaired Infant Lung Function with Sex-Specific Effects. Evidence from GRAPHS, a Cluster Randomized Cookstove Intervention Trial. Am J Respir Crit Care Med. 2019 Mar 15;199(6):738-746. doi: 10.1164/rccm.201804-0694OC. PMID 30256656
- [Derived] Quinn AK, Ae-Ngibise KA, Kinney PL, Kaali S, Wylie BJ, Boamah E, Shimbo D, Agyei O, Chillrud SN, Mujtaba M, Schwartz JE, Abdalla M, Owusu-Agyei S, Jack DW, Asante KP. Ambulatory monitoring demonstrates an acute association between cookstove-related carbon monoxide and blood pressure in a Ghanaian cohort. Environ Health. 2017 Jul 21;16(1):76. doi: 10.1186/s12940-017-0282-9. PMID 28732501
- [Derived] Jack DW, Asante KP, Wylie BJ, Chillrud SN, Whyatt RM, Ae-Ngibise KA, Quinn AK, Yawson AK, Boamah EA, Agyei O, Mujtaba M, Kaali S, Kinney P, Owusu-Agyei S. Ghana randomized air pollution and health study (GRAPHS): study protocol for a randomized controlled trial. Trials. 2015 Sep 22;16:420. doi: 10.1186/s13063-015-0930-8. PMID 26395578
- [Derived] Boamah EA, Asante K, Ae-Ngibise K, Kinney PL, Jack DW, Manu G, Azindow IT, Owusu-Agyei S, Wylie BJ. Gestational Age Assessment in the Ghana Randomized Air Pollution and Health Study (GRAPHS): Ultrasound Capacity Building, Fetal Biometry Protocol Development, and Ongoing Quality Control. JMIR Res Protoc. 2014 Dec 18;3(4):e77. doi: 10.2196/resprot.3797. PMID 25525828